CLINICAL TRIAL: NCT06523036
Title: Integrating Chiropractic Care and Mind-Body Training for the Treatment of Nonspecific Chronic Neck Pain in Nurses
Brief Title: Integrating Chiropractic Care and Mind-Body Training for the Treatment of Nonspecific Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Peter M. Wayne, Ph.D., Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019P003845
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Neck Pain; Nurse-Patient Relations
Keywords: Chiropractic; Tai Chi; Integrative Medicine
MeSH Terms: conditions — Neck Pain | interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined chiropractic care and Tai Chi (Experimental): All participants will be enrolled in a 16-week intervention period during which time they will receive 10 chiropractic treatments in addition to weekly Tai Chi training.
  Interventions: Procedure: Combined chiropractic care and Tai Chi

INTERVENTIONS:
Procedure: Combined chiropractic care and Tai Chi — Chiropractic will be personalized to the patients clinical needs within the scope of chiropractic practice in the Commonwealth of Massachusetts including: posture correction/spinal stabilization exercises; soft tissue relaxation techniques; spinal manipulation/mobilization; breathing and relaxation techniques; stretches, self-care; ergonomic modifications; bracing and supports. Chiropractic will be administered by one of two chiropractors at the Osher Clinical Center. Tai Chi will take place at one of two schools used in prior NIH funded trials.

SUMMARY:
Chronic neck pain is particularly prevalent among nurses. Nurses experiencing neck pain frequently report its impacts including decreased job satisfaction and reduced productivity. In recent years, non-pharmacologic approaches have increasingly been used treatments for the management of neck pain. Exercise and manual therapies represent two of the most common non-pharmacologic interventions for pain. The purpose of this study was to perform a pilot study of combined multimodal chiropractic care and Tai Chi for neck pain in nurses to help inform the design of a future, full-scale pragmatic trial.

DETAILED DESCRIPTION:
The lifetime prevalence of chronic neck pain is approximately 50%, and it is associated with substantial societal and individual burden. Neck pain is prevalent among healthcare workers, specifically among nurses. About 45% of nurses experience neck pain, but rates may vary by population and nursing type. Neck pain in nurses significantly contributes to sickness absence and negatively impacts nurses' productivity and performance at work. Neck pain is a burden on nurses' individual health and on the healthcare system as a whole. Two of the most common non-pharmacological approaches for the management of neck pain are exercise and manual therapies, and there is some evidence that multimodal approaches combining the two are more effective than unimodal strategies. Given the widespread availability in most metropolitan areas of both Tai Chi and chiropractic care, development of an evidence-based care regimen integrating Tai Chi mind-body self-care with chiropractic represents a practical strategy for management of neck pain.

To help inform the design of a larger-scale trial evaluating the combined effects of Tai Chi and chiropractic care for neck pain, the investigators propose to conduct a single-arm pilot study to evaluate the feasibility of delivering coordinated chiropractic care and Tai Chi via community-practitioners for nurses at Mass General Brigham Hospitals with chronic neck pain. 21 nurses with chronic neck pain that meet all study eligibility criteria will be recruited to receive 10 chiropractic treatments and weekly Tai Chi training over 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Nurses employed at Mass General Brigham Hospitals
* Chronic nonspecific neck pain at least 5 days a week for at least 3 consecutive months
* Neck pain level of 3 or higher as reported on a numerical scale ranging from 0 to 10, with 10 described as 'worst neck pain imaginable'
* Agreeable to participate and commit to study interventions
* Neck Disability Index score of 5 or greater
* Fluent in English

Exclusion Criteria:

* Currently, or having received chiropractic care in past 12 months
* Regular practice (on average, weekly) of Yoga, Tai Chi or Qigong in the past 6 months
* Any major systemic illness or unstable medical or psychiatric condition requiring immediate treatment or that could lead to difficulty complying with the protocol
* Any disability precluding exercise practice
* History of stroke, carotid artery dissection, or vertebral artery dissection
* Signs of myelopathy or carotid bruits or evidence of pathological hypermobility (e.g. Ehlers Danlos Syndrome) during the clinical exam
* Neck pain caused by congenital deformity of the spine that contraindicate treatment, neck pain related to neoplasm, inflammatory rheumatic disease, neurological disorder, active oncologic disease, severe affective disorder, addiction, or psychosis
* Neck pain associated with radicular pain or radiculopathy
* Pregnancy
* Recent spinal injections (in the past 4 weeks)
* Neck pain with litigation, any prior cervical surgery/spinal surgery within previous year
* Persons currently involved in a disability/accident claim

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Recruitment | 6 months
  Rate of enrollment (number of interested participants/number enrolled) and the percentage of eligible participants who consented to participate.
Retention | 16 weeks
  Percentage of participants who completed the 16-week intervention and follow-up measures.
Adherence to interventions | 16 weeks
  Proportion of participants who attend 70% of the chiropractic visits and 60% of the weekly Tai Chi classes.

SECONDARY OUTCOMES:
Pain Severity | Assessed at baseline and at week 16.
  Measured using a 11-point numerical rating scale (NRS) with 0 indicating "no pain at all" and 10 indicating "worst neck pain imaginable".
Neck Disability Index (NDI) | Assessed at baseline and at week 16.
  Self-report questionnaire used to determine how neck pain impacts daily activities of living and self-related neck pain disability. Scores range from 10 - 60. Higher scores indicate greater disability.
Pain on Movement (POM) | Assessed at baseline and at week 16.
  Participants are asked to flex, extend, laterally flex, and laterally rotate their necks to the left and right. The evoked pain is measured on a 11-point numerical rating scale (NRS) with 0 indicating "no pain at all" and 10 indicating "worst neck pain imaginable", for each direction. An average score is taken, with scores closer to 10 indicating more pain.
Bothersomeness of Pain | Assessed at baseline and at week 16.
  Measured using a 11-point numerical rating scale (NRS) with 0 indicating "neck pain not at all bothersome" and 10 indicating "neck pain extremely bothersome".
Patient Reported Outcome Measures Information System 29 (PROMIS-29) | Assessed at baseline and at week 16.
  A system of validated, highly reliable self-reported measures of health status for physical, mental, and social well-being. Raw scores are rescaled to standardized T-scores with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the item being measured.
Maslach Burnout Inventory (MBI) | Assessed at baseline and at week 16.
  A 3-section, 22-item self-report introspective psychological inventory pertaining to occupational burnout. Raw scores for the first subscale range from 0-54, for the second range from 0-30, and for the third range from 0-48. A higher score in the first two sections and a low score in the last section may indicate the presence of burnout.
Generalized Self-Efficacy Scale (GSES) | Assessed at baseline and at week 16.
  The GSES consists of 10 items with a 4-point Likert response scale ranging from 1 ("not at all true") to 4 ("exactly true"). Higher summed scores indicate greater self-efficacy to complete the task.
Hospital Anxiety and Depression Scale | Assessed at baseline and at week 16.
  A 14-item self-report questionnaire, with two seven-item sub scales, that measures current feelings of anxiety and depression. The total score for each sub scale ranges from 0-21, with higher scores representing higher levels of depression and anxiety.
Multidimensional Assessment of Interoceptive Awareness (MAIA) | Assessed at baseline and at week 16.
  A self-report questionnaire consisting of 8 scales, addressing 5 dimensions of body awareness. Dimensions are scored individually, and scores for each question are between 0-5, where higher scores equate to more awareness of bodily sensation.
Tampa Scale for Kinesiophobia | Assessed at baseline and at week 16.
  A 17-item self-report instrument that measures pain-related fear. Scores range from 17-68, with higher scores indicating higher levels of kinesiophobia.
Stanford Presenteeism Scale, 6-item version (SPS-6) | Assessed at baseline and at week 16.
  SPS-6 is a 6-item questionnaire assessing work quality and productivity. Scores range from 6-30, with higher scores indicating increased presenteeism.
Trail Making Test II | Assessed at baseline and at week 16.
  This two part cognitive tests is scored based on the number of sections it takes to complete each part of the test. Scores higher than the population average indicate higher degrees of cognitive impairment.
Gait Speed | Assessed at baseline and at week 16.
  Will be assessed using the ZenoTM Walkway, developed by ProtoKinetics (https://www.protokinetics.com). Participants will be asked to complete walking trials under a quiet walking condition, a fast-speed walking condition, and while completing a cognitive dual task.
Postural Awareness Scale | Assessed at baseline and at week 16.
  This 12-item self-report scale includes items that describe the awareness of body posture and postural control. Scores range from 12-84, with higher scores indicating greater postural awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- Osher Center for Integrative Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Given the pilot nature of this study, de-identified aggregate data will be shared in the dissemination of the main trial findings. As done with other trials in the Division of Preventive Medicine at Brigham and Women's Hospital, new research collaborations will be encouraged that make use of the data collected during this trial. Investigators interested in using data from this trial will be directed to contact the multiple principle investigators for data access.
  At all times, we are fully cognizant of and will scrupulously follow the guidelines of the Health Insurance Portability and Accountability Act (HIPAA), to ensure that participants' rights and confidentiality are not compromised.

REFERENCES:
- [Derived] Burton W, Wayne PM, Litrownik D, Long CR, Vining R, Rist P, Kilgore K, Lisi A, Kowalski MH. Integrating Chiropractic Care and Tai Chi Training for the Treatment of Chronic Nonspecific Neck Pain in Nurses: A Single-Arm Mixed-Methods Pilot Trial. J Integr Complement Med. 2024 Dec;30(12):1189-1199. doi: 10.1089/jicm.2024.0043. Epub 2024 Aug 22. PMID 39169834